CLINICAL TRIAL: NCT06511739
Title: A Phase 2 Randomized Double-blind Placebo-controlled Study to Evaluate the Efficacy and Safety of SYHX1901 Tablet in Non-segmental Vitiligo Patients
Brief Title: A Study to Evaluate the Efficacy and Safety of SYHX1901 Tablet in Non-segmental Vitiligo Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Collaborators: Zhongqi Pharmaceutical Technology (Shijiazhuang) Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYHX1902-004
Record Dates: First submitted 2024-07-02; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Non-segmental Vitiligo

STUDY DESIGN:
Intervention Model Description: Parallel assigned
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SYHX1901-A (Experimental): Participants in this group will receive dose A of SYHX1901 orally once daily (QD) for 52 weeks
  Interventions: Drug: SYHX1901
- SYHX1901-B (Experimental): Participants in this group will receive dose B of SYHX1901 orally QD for 52 weeks
  Interventions: Drug: SYHX1901
- SYHX1901-C (Experimental): articipants in this group will receive dose C of SYHX1901 orally QD for 52 weeks
  Interventions: Drug: SYHX1901
- Placebo followed by dose C of SYHX1901 (Placebo Comparator): Participants in this group will receive placebo orally QD for 24 weeks followed by dose C of SYHX1901 orally QD for 28 weeks.
  Interventions: Drug: SYHX1901; Drug: placebo

INTERVENTIONS:
Drug: SYHX1901 — SYHX1901 tablet
Drug: placebo — Oral tablet
  Arms: Placebo followed by dose C of SYHX1901

SUMMARY:
A 52-Week Study of SYHX1901 tablet in Adults with non-segmental vitiligo.

DETAILED DESCRIPTION:
SYHX1901 tablet is being evaluated for the treatment of non-segmental vitiligo. The study will enroll approximately 144 participants aged 18-65 with non-segmental vitiligo in 4 treatment arms. Participants will either receive study drug vs placebo oral tablets once daily (QD) for 24 weeks (Period A). In Period B (up to 52 weeks), participants who received placebo during the first 24 weeks will switch to study drug. Participants who received study drug during the first 24 weeks, will continue to receive study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign an ICF, able to comprehend and comply with the study procedures.
2. Male or female subjects aged 18 to 65，inclusive.
3. Subjects with a clinical diagnosis of non-segmental vitiligo.
4. Agree to stop all other treatments for vitiligo during the study period.
5. Women of child-bearing potential must have a negative serum pregnancy test within 3 days prior to the first study agent administration.

Exclusion Criteria:

1. Diagnosed as other active depigmentation disease.
2. At screening or baseline visits, subject exhibits active inflammatory dermatologic disease or symptoms that in the opinion of investigators would interfere of vitiligo evaluation or response to treatment.
3. Uncontrolled thyroid function at screening as determined by the investigator.
4. Use of permanent depigmentation treatment or skin grafts.
5. Use of phototherapy, topical or systemic treatments within certain time frame prior to Day1.
6. Have active bacterial/virus/other pathogens infection or infestation that require medical intervention.
7. Have progressive or uncontrolled systemic disease, or other concomitant chronic disease that the investigators believe unsuitable to participate the study.
8. History of alcohol and drug abuse within one year prior to screening; History of neurological or mental disorders with diagnosis records, such as severe depression, suicidal tendencies, epilepsy, dementia, etc.
9. Have any other reasons determined by the investigator that the subject is not eligible for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Facial-Vitiligo Area Scoring Index (F-VASI) | At 24 weeks
  The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.5.

SECONDARY OUTCOMES:
Percentage of Participants Achieving F-VASI 50 (≥ 50% Improvement in F-VASI From Baseline) | At 4、8、12、16、20、24、28、32、36、40、44、48、52、56 weeks
  The VASI is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.5.
Percentage of Participants Achieving F-VASI 75 (≥ 75% Improvement in F-VASI From Baseline) | At 4、8、12、16、20、24、28、32、36、40、44、48、52、56 weeks
  The VASI is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3.5.
Percentage of Participants Achieving Total Vitiligo Area Scoring Index (T-VASI) 50 (≥ 50% Improvement in T-VASI From Baseline) | At 4、8、12、16、20、24、28、32、36、40、44、48、52、56 weeks
  The VASI is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100.
Percent Change From Baseline in F-VASI | At 4、8、12、16、20、24、28、32、36、40、44、48、52、56 weeks
  The VASI is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100.
Percent Change From Baseline in BSA | At 4、8、12、16、20、24、28、32、36、40、44、48、52、56 weeks
  The BSA is measured by the number of hand units (palm plus 5 digits = 1% body surface area).
Change from baseline in Overall Dermatology Life Quality Index (DLQI) score | At 8、16、24、32、40、48、52、56 weeks
  The DLQI is a validated questionnaire used in dermatology clinical trials as patient reported outcome measure. The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week.
Change from baseline in Hospital Anxiety and Depression Scale (HADS) score | At 8、16、24、32、40、48、52、56 weeks
  The HADS is a self-rating patient reported outcome measure (PROM) to assess depression and anxiety in patients. Fourteen items are equally divided in two subscales: anxiety (HADS-A) and depression (HADS-D).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, China